CLINICAL TRIAL: NCT02086526
Title: Targeting Pathophysiologic Pathways in Polycystic Ovary Syndrome Using a Response to Metformin Phenotype
Brief Title: Targeting Pathways in Polycystic Ovary Syndrome (PCOS) Using Metformin (MET)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Alice Y Chang, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-000692; UL1TR000135 (NIH)
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin (Experimental): Metformin 500 mg. extended release (taken orally) one tablet with evening meal for one week, one tablet with morning and evening meal for one week, and one tablet at all three meals for the next three months.
  Interventions: Drug: Metformin
- Delayed Start Metformin (Other): After baseline study visit, this arm will return after three months without metformin for a repeat of the baseline study visit prior to initiating metformin 500 mg. extended release (taken orally) one tablet with evening meal for one week, one tablet with morning and evening meal for one week, and one tablet at all three meals for the next three months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Approximately 37 patients will start metformin therapy 3 months after their visit 2. All other patients will receive metformin therapy at their visit 2.
  Other Names: Glucophage, Glucophage XR, Glumetza, Fortamet, Riomet

SUMMARY:
The investigator's global hypothesis is that women with Polycystic Ovary Syndrome (PCOS) can be separated into subtypes based on their response to metformin. The investigators propose here to use both targeted and non-targeted metabolomic approach to identify pathways associated with metformin's effect on insulin sensitivity and endothelial function. This pilot project will be the foundation for developing tailored therapeutic approaches to Polycystic Ovary Syndrome and identifying novel drug targets.

DETAILED DESCRIPTION:
The investigators propose to use both targeted and non-targeted metabolomic approaches to identify pathways associated with metformin's effect on insulin sensitivity, weight, androgens and endothelial function. This project will be the foundation for developing tailored therapeutic approaches to Polycystic Ovary Syndrome and identifying novel drug targets. This pilot project is intended to inform the development of hypothesis and specific aims for a future grant application to National Institutes of Health (NIH).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 25
* Polycystic Ovary Syndrome criteria of both oligomenorrhea (<9 menses per year) and androgen excess [clinical hirsutism (Ferriman-Gallway score >8 or severe acne) or elevated testosterone].
* Taking no medications for the treatment of insulin resistance.

Exclusion Criteria:

* Diagnosis of Cushing's syndrome
* Untreated hypo/hyperthyroidism
* Elevated prolactin
* Congenital adrenal hyperplasia
* Renal insufficiency (creatinine > 1.5)
* Diabetes
* Medications that can significantly affect endothelial function
* Pregnancy
* Breast Feeding
* Taking oral contraceptives
* Currently smoking

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-03; Primary Completion 2016-11-20 (Actual); Study Completion 2016-11-20 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity (SI) after 3 Months of Metformin Therapy | Baseline, 3 months
  Insulin sensitivity will be calculated using an oral glucose minimal model. Insulin under the curve will be calculated geometrically with the trapezoidal rule.

SECONDARY OUTCOMES:
Change in Peripheral Flow-Mediated Vasodilatation after 3 Months of Metformin Therapy | baseline, 3 months
  The ratio of Peripheral Digital Arterial Tonometry (PAT) signal after cuff release compared with baseline is calculated through a computer algorithm normalizing for baseline measurements and indexing to measurements in the contra-lateral arm. The calculated ratio reflects the reactive hyperemia index (RHI).

OTHER OUTCOMES:
Change in Weight | baseline, 3 months
Change in Testosterone | baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alice Chang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Heidari B, Lerman A, Lalia AZ, Lerman LO, Chang AY. Effect of Metformin on Microvascular Endothelial Function in Polycystic Ovary Syndrome. Mayo Clin Proc. 2019 Dec;94(12):2455-2466. doi: 10.1016/j.mayocp.2019.06.015. PMID 31806099